CLINICAL TRIAL: NCT00968396
Title: Ex-Vivo Depletion of Myeloma Cells From Peripheral Blood Progenitor Cell Grafts
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0886
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Ex-Vivo Depletion of Myeloma Cells; Peripheral Blood Progenitor Cell Grafts; PBPC; Stem Cell Transplant; Bone marrow stem cells; Melphalan; Alkeran; Apheresis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Blood Component Removal; Stem Cell Transplantation; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cell Collection + Transplantation (Experimental): Apheresis: On Day 5, 3 hour process to separate blood (stem cells from other cells) done 1 time a day for 1-6 days, or until enough stem cells are collected. Stem cells are cultured with donated stem cells from a relative for two weeks before being returned via transplantation. Co-culture Stem Cell Infusion on Day 0. Melphalan 100 mg/m^2 IV over 30 minutes daily on Days -2 and -1.
  Interventions: Procedure: Apheresis; Procedure: Stem Cell Transplantation; Drug: Melphalan

INTERVENTIONS:
Procedure: Apheresis — On Day 5, 3 hour process to separate blood (stem cells from other cells) done 1 time a day for 1-6 days, or until enough stem cells are collected. Stem cells are cultured with donated stem cells from a relative for two weeks before being returned via transplantation.
Procedure: Stem Cell Transplantation — Co-culture Stem Cell Infusion on Day 0.
Drug: Melphalan — 100 mg/m^2 IV over 30 minutes daily on Days -2 and -1
  Other Names: Alkeran

SUMMARY:
The goal of this clinical research study is to learn if cleaning the stem cells of a patient who has multiple myeloma (MM) with the bone marrow of a relative will make a cell product capable of replacing the bone marrow after standard treatment with chemotherapy.

DETAILED DESCRIPTION:
A transplant of one's own bone marrow stem cells is part of a standard treatment for MM. Because MM comes from the bone marrow, stem-cell products from the bone marrow can have tumor cells mixed in them when they are transplanted. This may cause the disease to return after transplant. This study will learn about a method of cleaning, or "purging," the MM tumor cells from the stem cells by using the bone marrow of a relative.

Study Drugs:

Melphalan is designed to damage the DNA (the genetic material) of cells, which may cause cancer cells to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will be given G-CSF twice a day through a needle under the skin on Days 1-5 to move stem cells from out of the bone marrow and into the blood.

You will receive melphalan through a needle in your vein over 30 minutes each time on the 2 days directly before you receive the stem cell transplant.

Stem Cell Collection, Purging, and Transplantation:

On Day 5, stem cell collection will begin. You will have a central venous catheter (CVC - a sterile, flexible tube) placed into a vein in your chest while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

Blood will be removed from your body through the CVC and passed through a machine that separates stem cells from the other cells. The stem cells will be frozen for storage, and the blood will be returned to your body. This 3-hour process is called apheresis. This process will be done 1 time a day for 1-6 days, or until enough stem cells are collected.

Your stem cells will be placed in a sterile container, where they will grow and multiply with donated stem cells from a relative. If there are enough cells after 2 weeks, the cells will be transplanted back into the body. If there are not enough cells after the 2 weeks of growing with the donor's stem cells, they will be combined with a sample that was set aside at your initial collection and then transplanted back into the body.

Study Visits:

One (1), 2, and 6 months after the transplant, blood (about 2 teaspoons) will be drawn for routine tests and to check the status of the disease.

Six (6) months after the transplant, you will also have a bone marrow aspirate/biopsy to check the status of the disease.

Length of Study:

You will remain on study until 12 months after the transplant. You will be taken off study if the disease gets worse or needs further treatment.

End-of-Treatment Visit:

Twelve (12) months after the transplant, you will have your end-of-treatment visit. At this time, the following tests and procedures will be performed:

* Blood (about 2 teaspoons) will be drawn for routine tests and to check the status of the disease.
* You will have a bone marrow aspirate/biopsy.
* You will have x-rays taken of your bones.

This is an investigational study. Melphalan is FDA approved and commercially available for the treatment of MM. While receiving a stem-cell transplant is standard treatment for MM, cleaning (purging) the stem-cell product is investigational.

Up to 25 recipients will take part in this study. All will be enrolled at M. D. Anderson

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple myeloma who have relapsed after an autologous transplant or with a chemosensitive relapse more than one year post initial therapy
2. Age 18 to 75 years
3. Left ventricular ejection fraction >/= 40%. No uncontrolled arrhythmias
4. FEV1, FVC and DLCO >/= 40%. No symptomatic pulmonary disease
5. Serum bilirubin </= 2 x upper limit of normal, SGPT </= 4 x upper limit of normal
6. HIV-negative
7. Negative Beta HCG test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization
8. Patient or guardian able to sign informed consent
9. Marrow-MSC Donor Requirements: patients must have a family member who is matched at 2, 3, or 4 HLA antigens and willing to donate 80-100 ml or bone marrow for MSC generation

Exclusion Criteria:

1. International Staging System (ISS) stage I at diagnosis (beta-2 microglobulin < 3.5 mg/L and albumin >/= 3.5 g/dL)
2. Patients with an apheresis collection </= 7 x 10e6 CD34+/Kg
3. A fully matched related donor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Neutrophil Engraftment Rate | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Yago Nieto, MD, PHD, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org